CLINICAL TRIAL: NCT05451784
Title: Treatment of Advanced or Metastatic Triple-negative Breast Cancer With Adoptive Therapy of PD1+ Tumor-infiltrating Lymphocytes (TILS001 Trial)
Brief Title: Treatment of Advanced or Metastatic Triple-negative Breast Cancer With Adoptive Therapy of PD1+ TILS
Acronym: TILS001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacio Clinic Barcelona (Other)
Collaborators: SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILS001 trial
Record Dates: First submitted 2022-07-04; First posted 2022-07-11 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Triple-Negative Breast Carcinoma
Keywords: TNBC; Breast Cancer; metastatic; triple negative
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD1+ TILs (NUMARZU-001) product infusion (Experimental): The treatment administration is divided in NMA-LD chemotherapy(auxiliary medication), TILs product (IMP) and IL-2 (auxiliary medication).
  Interventions: Drug: PD1+ TILs (NUMARZU-001) product infusion

INTERVENTIONS:
Drug: PD1+ TILs (NUMARZU-001) product infusion — The cryopreserved NUMARZU-001 product will be thawed in a 37ºC water bath and will be infused by gravity, a 5 mL to 10 mL/ minute.
  Concomitant medications will be given to the patient starting within 24 hours before NUMARZU-001 product infusion. This therapy will include the following:
  * Hydration as per institutional standards (Saline solution 0,9% NaCl 500ml every 8 hours) 24 hours before the NUMARZU-001 product infusion.
  * Within 30 to 60 minutes before infusion of NUMARZU-001, premedicate the patient with paracetamol (1 g) and dexclorfeniramina (5 mg IV), or another H1- histamine antagonist.
  Continuous supervision of the patient by site medical staff is required until completion of infusionof the NUMARZU-001 product, to monitor for potential signs and symptoms (e.g. hypersensitivityreaction).
  Other Names: TILs

SUMMARY:
This is a prospective, multicenter, phase I/II, open-label, two-stage design of PD1+ TILs infusion in metastatic or advanced TNBC. TILS001 includes 3 parts. Previous to each phase inclusion, a specific ICF must be signed by the patient. Participants potentially eligible to participate in the clinical trial will be offered to sign a ICF three times prior to TILs treatment: 1) to allow for collection of archival FFPE tissue samples for determination PD1 by mRNA (Part #1), 2) prior to a fresh metastatic biopsy for selection, isolation and partial expansion of PD1+ TILs (Part #2) and 3) prior to allow for remaining study procedures and TILs therapy (Part #3, Main Consent).

DETAILED DESCRIPTION:
This trial has been developed in TNBC, a breast cancer subtype with a particularly poor prognosis. The product used for treating participating patients will be selected PD1-positive TILs. Such TILs will be manufactured in Hospital Clinic under the name of NUMARZU-001. The procotol has been designed in three parts to better select participating patients. Molecular pre-screening has been established to select tumors with a higher probability of enrichment by PD1-positive TILs. The pre- screening consists of performing a tumor biopsy and selecting isolation and expansion of PD1- postive TILs to manufacture the final product NUMARZU-001. This part could last almost four weeks, as such patients will continue with the established treatment in the meanwhile. Finally, NUMARZU-001 will be administered if the patient is eligible for part three of the protocol.

ELIGIBILITY:
Eligibility criteria for Part #1 (Molecular pre-screening: Determination of PD1 by mRNA analysis from an archival FFPE tumor sample):

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Age ≥ 18 years.
2. Estimated life expectancy of ≥6 months.
3. Histologically confirmed diagnosis of unresectable or metastatic breast cancer.
4. Histologically confirmed diagnosis of advanced triple-negative breast cancer (based on the most recently analyzed biopsy from locally recurrent or metastatic site, local laboratory) meeting the following criteria: HER2-negative in situ hybridization test or an immunohistochemistry (IHC) status of 0 or 1+, and ER and PgR expressions <10% as determined locally by IHC assay as per most recent ASCO/CAP guidelines.
5. Patients could have received a maximum of 5 lines of prior standard of care chemotherapy in the inoperable/metastatic setting.
6. Patients must not have history of other malignancy within the past 3 years with the following exceptions: adequately treated non-melanoma skin cancer without evidence of disease at the time of enrollment; adequately treated cervical carcinoma in situ without evidence of disease at the time of enrollment; adequately treated breast ductal carcinoma in situ without evidence of disease at the time of enrollment; prostatic intraepithelial neoplasia without evidence of prostate cancer at the time of enrollment; adequately treated superficial or in-situ carcinoma of the bladder without evidence of disease at the time of enrollment.
7. Subject likely to be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
8. Absence of psychiatric or physiologic history, substance abuse, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
9. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
10. Pregnant or breastfeeding women will NOT be eligible.
11. Subject has known sensitivity to any of the products or components to be administered during dosing will NOT be eligible.
12. NOT having an immediate family member (eg, spouse, parent/legal guardian, sibling, or child) who is investigational site or sponsor staff directly involved in this trial, unless prospective institutional review board (IRB)/independent ethics committee (IEC) approval (by chair or designee) is given allowing an exception to this criterion for a specific subject
13. Patients must NOT have undergone prior allogeneic hematopoietic stem cell transplantation
14. Patients with a history or evidence of symptomatic autoimmune will NOT be eligible: glomerulonephritis, vasculitis, or other symptomatic autoimmune diseases, or active autoimmune disease or syndrome that has required systemic treatment in the past 2 years (ie, with the use of disease-modifying agents, corticosteroids or immunosuppressive drugs) except vitiligo or resolved childhood asthma/atopy. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Absence of active bacillus tuberculosis history.
16. Absence of a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required.
17. Absence of a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required.
18. To be able to provide either a newly obtained tumor biopsy (preferred) or archival tumor tissue of an FFPE tumor block. The tumor tissue should be of good quality based on total and viable tumor content and must be evaluated centrally for gene expression analysis prior to enrollment in Part #2.

Eligibility criteria for Part #2 (Pre-Screening Phase: Selection, isolation and partial expansion of PD1+ TILs from a fresh tumor sample):

Participants are eligible to be included in the study only if all the previous and the following criteria apply:

1. Patients will be eligible for Part #2 if they have a PD-1 mRNA expression above the 20th percentile in the FFPE tumor sample analyzed in Part 1.
2. At least 1 resectable target lesion
3. Patients must NOT have clinically active cerebral metastases. Carcinomatous meningitis is not allowed regardless of clinical stability.

Eligibility criteria for Part #3 (Screening and treatment Phase: Complete expansion of PD1+TILs. Treatment of patients with PD1+ TILs infusion):

Participants are eligible to be included in the study only if all of the previous and the following criteria apply. For being included in this section, the following criteria must apply:

1. PD1+ TILs selection in Part #1 and successful partial expansion of tumor sample in Part #2
2. Treatment-related toxicities (except alopecia and neuropathy G2) must ≤ Grade 1 at the time of allocation according to CTCAE version 5.0.
3. All patients must have received two or more prior systemic therapies, including at least one of them for advanced disease and an ADC. A maximum of five chemotherapy-based lines are permitted in the metastatic setting. Prior treatment should be discontinued 28 days or 5 half-lives, whichever is shorter, before day 1 of NMA-LD.
4. Measurable disease according to RECIST 1.1 criteria.
5. Adequate organ function determined within 28 days prior to enrollment.
6. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to enrollment.
7. For patients ≥ 60 years or patients who have a history of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias, a cardiac stress tests must be performed showing normal LVEF, NYHA functional classification < class 1 and if any wall movement abnormalities, they must be reversible.
8. Left ventricular ejection fraction (LVEF) ≥ 50% at baseline as determined by either ECHO or MUGA
9. Patients must not be currently receiving treatment with another investigational device or drug study. No other investigational procedures (of any kind) are permitted while participating in this study.
10. Systemic steroid therapy is not permitted (patients who require replacement therapy for adrenal insufficiency may be enrolled if the steroid treatment dose does not exceed 10 mg of prednisone or equivalent).
11. Patients with evidence of clinically significant immunosuppression will NOT be eligible.
12. Patients with evidence of (non-infectious) pneumonitis that required steroids or current pneumonitis will NOT be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3-5 adverse event (AE) | 24 weeks from the administration of PD1+ TILS (NUMARZU-001 product)
  Incidence of grade 3-5 adverse event (AE) assessed by the NCI Common Terminology for Classification of Adverse Events (CTCAE) version 5.0, and any grade AE assessed by CTCAE that leads to treatment discontinuation and possibly related to treatment, that occur in the first 24h following PD1+ TILs infusion (prior to IL-2 treatment).
  * Incidence of grade 3-5 AEs assessed by the NCI CTCAE version 5.0 taking into account the whole process, which includes NMA-LD chemotherapy followed by TILs infusion and at least one dose of IL-2 treatment.
  * All changes in treatment administration including delays, interruptions, reductions or discontinuation and the main reason(s) for these changes.
Overall response rate (ORR) | 24 weeks from the administration of PD1+ TILS (NUMARZU-001 product)
  Overall response rate (ORR) locally determined as the best response (defined as CR and PR) by the investigator according to RECIST 1.1 criteria from the administration of PD1+ TILS (NUMARZU-001 product); on day 0

SECONDARY OUTCOMES:
Progression-Free Survival at 6 months(PFS6) | 24 weeks from the administration of PD1+ TILS (NUMARZU-001 product)
  Progression-Free Survival at 6 months(PFS6) defined as the proportion of patients alive and without progression (as determined locally by the investigator according to Response Evaluation Criteria in Solid Tumor [RECIST] 1.1 version) 24 weeks from the administration of PD1+ TILS (NUMARZU-001 product); on day 0
Clinical Benefit Rate at 6 months (CBR6) | 24 weeks from the administration of PD1+ TILS (NUMARZU-001 product)
  Clinical Benefit Rate at 6 months (CBR6) from the administration of PD1+ TILS (NUMARZU-001 product); on day 0 defined as Complete response (CR), Partial response (PR) or Stable Disease (SD) for at least 6 months, as determined locally by the investigator according to RECIST 1.1 criteria.
Duration of Response (DoR) | 24 weeks from the administration of PD1+ TILS (NUMARZU-001 product)
  Duration of Response (DoR) defined as the time from the first occurrence of a documented objective response to disease progression, as determined locally by the investigator using RECIST v1.1, or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | 24 weeks from the administration of PD1+ TILS (NUMARZU-001 product)
  Progression-free survival (PFS) defined as the timefrom the administration of PD1+ TILS (NUMARZU-001 product); on day 0 to the first occurrence of disease progression, as determined locally by the investigator using RECIST v1.1, or death due to any cause, whichever occurs first.
Overall Survival (OS) | From completion of the Response Assessment Period and up to 5 years from the last study treatment until death, loss to follow-up, or withdrawal of consent
  Overall Survival (OS) defined as the time from the administration of PD1+ TILS (NUMARZU-001 product); on day 0 to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Aleix Prat, Study Chair — Hospital Clinic; Laura Angelats, Study Chair — Hospital Clinic
Locations (4):
- Spain (4):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Clínica universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No